CLINICAL TRIAL: NCT07259772
Title: Anesthetic Effect of Ropivacaine on Local Infiltration Anesthesia in Arteriovenous Fistula Surgery: a Randomized Controlled Trial
Brief Title: Anesthetic Effect of Ropivacaine on Local Infiltration Anesthesia in Arteriovenous Fistula Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LW-20241021002-01
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: End Stage Renal Disease (ESRD); Arteriovenous Fistula Patency; Chronic Kidney Disease 5D
Keywords: Ropivacaine; Local Anesthesia; Infiltration Anesthesia; Arteriovenous Fistula Surgery; Hemodialysis Access; Randomized Controlled Trial; Vascular Access; Lidocaine; Pain Control
MeSH Terms: conditions — Kidney Failure, Chronic; Agnosia | interventions — Ropivacaine; Lidocaine

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel group randomized controlled trial comparing ropivacaine versus lidocaine for local infiltration anesthesia in arteriovenous fistula surgery. Participants are randomly assigned to one of two treatment groups and remain in that group throughout the study period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study where both patients and surgeons are blinded to the intervention. The anesthetic preparations are performed by resident physicians, circulating nurses, and scrub nurses who are not involved in outcomes assessment. The allocation assignments are concealed in sequentially numbered, opaque, sealed envelopes that are opened immediately prior to anesthesia administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine Group (Experimental): Patients receiving 0.375% ropivacaine (75 mg in 20 mL) for local infiltration anesthesia
  Interventions: Drug: Ropivacaine
- Lidocaine Group (Active Comparator): Patients receiving 0.67% lidocaine (100 mg in 15 mL) for local infiltration anesthesia
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Ropivacaine — 0.375% ropivacaine solution (75 mg total dose in 20 mL volume) administered as local infiltration anesthesia for arteriovenous fistula surgery
  Arms: Ropivacaine Group
Drug: Lidocaine — 0.67% lidocaine solution (100 mg total dose in 15 mL volume) administered as local infiltration anesthesia
  Arms: Lidocaine Group

SUMMARY:
This study compares two local anesthetics, ropivacaine and lidocaine, for patients undergoing arteriovenous fistula surgery. Arteriovenous fistula is the preferred vascular access for end-stage kidney disease patients needing hemodialysis.

In this clinical trial, patients are randomly assigned to receive either ropivacaine or lidocaine for local anesthesia during the surgery. Researchers are evaluating which medication provides better pain control and improves surgical outcomes.

The study is examining:

* Pain levels during and after surgery
* Surgery duration
* Need for additional pain medication
* Surgical complications
* Fistula development over time
* Long-term fistula function at 1 year and 5 years

This is a double-blind study, meaning neither patients nor surgeons know which medication is being used. The study is currently ongoing with active patient follow-up and is expected to be completed in June 2026. Patients are being followed for up to 5 years to monitor their long-term progress.

This research may help doctors choose the best local anesthetic for arteriovenous fistula surgery, potentially leading to better pain control and improved long-term outcomes for kidney disease patients.

DETAILED DESCRIPTION:
Blinding & Drug Preparation: To maintain blinding, all anesthetic solutions were prepared by the hospital pharmacy under aseptic conditions. Both solutions were clear, colorless, and dispensed in identical 20mL syringes labeled only with the study ID and patient randomization number.

Standardized Infiltration Protocol: A fixed sequence was used: subcutaneous infiltration along the planned 3-4 cm incision line, followed by targeted perivascular infiltration around the exposed radial artery and cephalic vein using a 25-gauge needle.

Standardized Surgical Protocol (Per Study Procedures): All surgeries were performed by the same high-volume surgeon. With the patient in the supine position and the operative limb abducted, a 3-4 cm skin incision was made between the artery and vein. The cephalic vein and radial artery were carefully dissected. The distal cephalic vein was ligated and divided. While an assistant compressed the cubital fossa, heparinized saline (5000 IU in 500 mL saline) was injected through the proximal vein to fully dilate the forearm cephalic vein. Vascular clamps were then applied to occlude the radial artery. Parallel longitudinal incisions (0.8-1 cm) were made in both vessels. The anastomosis was completed using continuous everting sutures on both the anterior and posterior walls. After clamp release and confirmation of fistula patency, the incision was closed in layers.

Intraoperative Adjuncts: All patients received the aforementioned irrigation with heparinized saline for venous dilation.

Protocol-Specified Additional Monitoring & Quality Assurance:

Extended Monitoring: Beyond pre-specified outcomes, the protocol mandated daily wound assessments for the first postoperative week and monitoring for signs of local anesthetic systemic toxicity (LAST) within 24 hours.

Data Quality Control: To minimize bias, a single, uniformly trained research assistant, blinded to group allocation, was responsible for collecting all intraoperative and postoperative data, including pain scores. Source data verification was performed for all primary outcome measures.

Study Progress Context (as of November 2025): Patient enrollment (n=40) and all surgical procedures were completed between April 2019 and February 2020. The study is currently in the long-term follow-up phase, tracking the 5-year primary unassisted patency endpoint. Blinding has been maintained throughout follow-up. Final data collection for the 5-year endpoint is anticipated by June 2026.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18 years) scheduled for primary radiocephalic arteriovenous fistula creation
* Diagnosed with end-stage renal disease requiring hemodialysis
* Willing and able to provide written informed consent

Exclusion Criteria:

1. History of arteriovenous fistula on the ipsilateral limb
2. Impaired communication abilities or inability to complete questionnaires due to language barriers, or missing essential data
3. Preoperative ultrasound findings of:

   * Radial or brachial artery diameter <1.8 mm
   * Cephalic vein diameter <2 mm at the wrist or <3 mm at the elbow (without tourniquet application)
4. Known allergy to local anesthetics (ropivacaine or lidocaine)
5. Coagulopathy or bleeding disorders
6. Local infection at the planned anesthesia or surgical site
7. Severe peripheral neuropathy or neurological disorders affecting upper limb function
8. Significant thrombosis or severe stenosis in the proximal major veins or central veins of the limb
9. Pregnancy or breastfeeding
10. Participation in another clinical trial within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Pain Scores | During surgery (at the end of the procedure)
  Pain intensity assessed using 10-point Visual Analog Scale (0 = no pain, 10 = worst pain imaginable)
Operative Time | During surgery
  Duration from skin incision to wound closure (minutes)
Need for Supplemental Anesthesia | During surgery
  Requirement for additional anesthetic doses due to patient-reported intolerable pain after initial infiltration
Postoperative Pain Scores | 24 hours postoperatively
  Pain intensity assessed using 10-point Visual Analog Scale
Incidence of Postoperative Vasospasm | 48 hours postoperatively
  Development of arteriovenous fistula tremor reduction or absence within 48 hours postoperatively

SECONDARY OUTCOMES:
Surgical Success Rate | Immediately after surgery
  Successful creation of functional arteriovenous fistula
Postoperative Complications | 24 hours postoperatively
  Incidence of hematoma or hemorrhage within 24 hours after surgery
Fistula Maturation at 8 Weeks | 8 weeks postoperatively
  Clinical maturation defined as easily palpable vein with straight segment >10 cm, adequate diameter, and well-palpable thrill; OR ultrasonographic maturation defined as outflow vein diameter >6 mm, depth <6 mm, and blood flow >500 mL/min
Primary Unassisted Patency at 1 Year | 1 year postoperatively
  Interval from access creation until first access occlusion or any intervention to maintain/restore patency
Primary Unassisted Patency at 5 Years | 5 years postoperatively
  Interval from access creation until first access occlusion or any intervention to maintain/restore patency

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhang, Principal Investigator — Lianyungang First People's Hospital
Locations (1):
- Lianyungang First People's Hospital, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in publications will be shared, including demographic data, baseline characteristics, primary and secondary outcome measures, and safety data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will become available 6 months after publication of the primary results and will be accessible for 5 years.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be directed to the corresponding author. Requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Budharapu A, Sinha R, Uppada UK, Subramanya Kumar AV. Ropivacaine: a new local anaesthetic agent in maxillofacial surgery. Br J Oral Maxillofac Surg. 2015 May;53(5):451-4. doi: 10.1016/j.bjoms.2015.02.021. Epub 2015 Mar 24. PMID 25818492
- [Background] Lok CE, Huber TS, Lee T, Shenoy S, Yevzlin AS, Abreo K, Allon M, Asif A, Astor BC, Glickman MH, Graham J, Moist LM, Rajan DK, Roberts C, Vachharajani TJ, Valentini RP; National Kidney Foundation. KDOQI Clinical Practice Guideline for Vascular Access: 2019 Update. Am J Kidney Dis. 2020 Apr;75(4 Suppl 2):S1-S164. doi: 10.1053/j.ajkd.2019.12.001. Epub 2020 Mar 12. PMID 32778223
- [Background] Schmidli J, Widmer MK, Basile C, de Donato G, Gallieni M, Gibbons CP, Haage P, Hamilton G, Hedin U, Kamper L, Lazarides MK, Lindsey B, Mestres G, Pegoraro M, Roy J, Setacci C, Shemesh D, Tordoir JHM, van Loon M, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Lindholt J, Naylor R, Vega de Ceniga M, Vermassen F, Verzini F, Esvs Guidelines Reviewers, Mohaupt M, Ricco JB, Roca-Tey R. Editor's Choice - Vascular Access: 2018 Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Jun;55(6):757-818. doi: 10.1016/j.ejvs.2018.02.001. Epub 2018 May 2. No abstract available. PMID 29730128

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT07259772/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT07259772/ICF_001.pdf